

# Clinical Evaluation of Biomedics 1 day Toric and MyDay® toric

Sponsor Study Code: EX-MKTG-146

Protocol Date: November, 2022

Sponsor Company: CooperVision, Inc.

Document Type: Protocol

Study Category: Post Market

Start Date: January, 10th 2023

Finish Date: March, 31 2023

Clinical Site: Clinic of Optometry, Faculty of Optics and

Optometry; Universidad Complutense de Madrid



#### **Revision History**

| Document number | Date | Comments |
|-----------------|------------|-----------------------|
| EX-MKTG-146 | 11/28/2022 | First draft (v 1.0) |
| EX-MKTG-146 | 11/29/2022 | First draft (v 2.0) |
| EX-MKTG-146 | 11/29/2022 | Final protocol (v3.0) |



# **Protocol Synopsis**

| Protocol Number | EX-MKTG-146 |
|---|---|
| Title | Clinical Evaluation of Biomedics 1 day Toric and MyDay® toric |
| Name of Device(s) and (by USAN material) | Biomedics 1 day toric (ocufilcon D), MyDay toric (stenfilcon A) |
| Indications for Use | Approved for use: |
| Study Design | Subject masked, interventional, prospective, direct refit, bilateral wear study. |
| Purpose | The aim of this non-dispensing fitting study is to evaluate the short term lens fit, vision performance and patient subjective experiences of the Biomedics 1 day toric when compared to the MyDay toric after 15 minutes of daily wear. |
| Study Duration | The anticipated timeline for this study is as follows: • Patient enrolment and completion: January - February 2023 Visits: V1: (BL/trial fit/lens order), V2: Dispense / evaluate P1 V3: 15 minutes. Evaluate P1/Dispense P2. V4: 15 minutes. Evaluate P2 / study exit |
| Patient Population | Habitual soft toric contact lens wearers who provide written informed consent and meet the protocol entrance criteria. |
| Sample Size | Target enrollment and completion is 37subjects. |
| Center Destination (Mexico) | Consultorio Optométrico Queretaro # 238-604 Colonia Roma,<br>Cuauhtémoc. Ciudad de México. Código Postal 06760 |
| Number of Centers | Single Center |
| Patient Follow-up | Subjects enrolled in this study will be followed up after the lens dispensing session: • Post dispensing follow-up at 15 minutes for each study lens pair |
| Primary Endpoint | Subjective handling (insertion & removal) |

### **Table of Contents**

| 1 | I | ntro | duction | 6 |
|---|---|---|---|---|
| 2 | S | Study | y Objective | 6 |
| 3 | S | Study | y Hypothesis | 6 |
| | 3.1 | 5 | Study Hypothesis | 6 |
| 4 | S | Study | y Design | 7 |
| 5 | I | nves | tigational Sites | 7 |
| | 5.1 | 1 | Number of Sites | 7 |
| | 5.2 | I | nvestigator Recruitment | 7 |
| 6 | E | Ethic | s Review / Statement of Compliance | 7 |
| | 6.1 | F | Relevant Standards / Guidelines | 7 |
| | 6.2 | I | nstitutional Review Board | 7 |
| | 6.3 | ( | Clinical Trial Registration | 7 |
| | 6.4 | I | nformed Consent | 8 |
| 7 | F | Poter | ntial Risks and Benefits to Human Subjects | 8 |
| 8 | N | /late | rials and Methods | 9 |
| | 8.1 | F | Participants | 9 |
| | li | nclus | sion criteria | 9 |
| | 8.2 | 5 | Study Materials | 10 |
| | 8 | 3.2.1 | Contact lens | 10 |
| | 8 | 3.2.2 | Contact Lens care | 11 |
| | 8 | 3.2.3 | Storage of Study Medications/Treatments | 11 |
| | 8 | 3.2.4 | Clinical Supply Inventory | 11 |
| | 8 | 3.2.5 | Disposal of Consumables | 11 |
| | 8 | 3.2.6 | Masking and Control of Study Materials | 11 |
| | 8 | 3.2.7 | Ordering and Accountability of Study Materials | 12 |
| | 8.3 | ١ | Visit Schedule and Procedures | 12 |
| | 8 | 3.3.1 | Visit 1: Baseline / Trial Fit / Lens order | 12 |
| | 8 | 3.3.2 | Visit 2: Lens dispensing (Fit LENS A / Evaluate) | 13 |
| | 8 | 3.3.3 | Visit 3: 15 minutes (Evaluate LENS A) | 13 |
| | 8 | 3.3.4 | Visit 3: Lens dispensing (Fit LENS B / Evaluate) | 13 |
| | 8 | 3.3.5 | Visit 4: 15 minutes (Evaluate LENS B / Study Exit) | 14 |
| C | onfide | ential | | 4 |

| 9 | Adv | verse Event Reporting | 14 |
|----|-------|--------------------------------|----|
| | 9.1 | Adverse Response Definitions | 14 |
| | 9.2 | Procedures for Adverse Events | 16 |
| | 9.3 | Reporting Adverse Events | 17 |
| | 9.4 | Discontinuation from the Study | 17 |
| 10 | ) Sta | tistical Analysis | 17 |
| | 10.1 | Statistical analysis | 17 |
| | 10.2 | Sample size | 18 |
| 11 | Dat | a Quality Assurance | 19 |
| | 11.1 | Study monitoring | 19 |
| | 11.2 | Record keeping | 19 |
| | 11.3 | Record retention | 19 |
| | 11.4 | Data Entry / Data Management | 19 |
| | 11.5 | Confidentiality | 19 |
| | 11.6 | Publication | 19 |
| 12 | 2 | | |

### 1 Introduction

A recent publication from 2021 comparing the data in the US market from three sources, indicates that the daily disposable modality continues to lead in terms of prescribing by soft lens replacement schedule (range of 43% to 51%)¹. Toric soft contact lenses, (TSCL), work best for people with astigmatism and other refractive errors (e.g., nearsightedness, farsightedness). The use of toric soft contact lenses (TSCL) has increased significantly in recent years. Soft toric contact lens wearers demand two things from their contact lenses, great comfort and excellent vision. Recently released data on prescription habits with soft toric lenses ranged from 13% to 59%. Contact lens manufacturers are continuously innovating in this area, with increased availability of soft toric contact lenses with novel designs in a range of replacement frequencies, from daily disposables to monthly replacement, and different materials, including silicone hydrogels.

Therefore, CooperVision is interested in comparing the short-term clinical performance and subjective acceptance of Biomedics 1 Day Toric hydrogel contact lenses (**LENS A**) with MyDay Toric (**LENS B**) silicone hydrogel lenses. A non-dispensing fitting study is proposed to evaluate the short-term clinical performance of these two daily disposable lenses.

## 2 Study Objective

The aim of this non-dispensing fitting study is to evaluate the short term lens fit, vision performance and patient subjective experiences of the Biomedics 1 Day Toric when compared to the MyDay Toric lenses after 15 minutes of daily wear.

#### The primary outcome variable is:

Subjective handling ratings on insertion (assessed by subjects)



## 3 Study Hypothesis

## 3.1 Study Hypothesis

- Null hypothesis (Ho): There is no difference in clinical performance and subjective assessments between toric lens types.
- Alternative hypothesis (H1): There is a difference in clinical performance and subjective assessments between toric lens types.

## 4 Study Design

This is a subject masked, interventional, prospective, direct refit, bilateral wear study. It is anticipated that this study will involve 4 visits as follows: **V1:** (BL/trial fit/lens order), **V2:** Dispense / evaluate P1. **V3:** 15 minutes. Evaluate P1/Dispense P2. **V4:** 15 minutes. Evaluate P2 / study exit.

## 5 Investigational Sites

#### 5.1 Number of Sites

This will be a single center investigational site in Madrid (Spain) (Target 40 subjects).

## 5.2 Investigator Recruitment

This study was conducted at School of Optometry Clinic; at the University Complutense of Madrid (Spain). The Investigators will be required to fulfil the following criteria:

- Licensed optometrist with at least two years of contact lens fitting experience.
- Experienced Investigators who will be trained in Good Clinical Practice (GCP) by the principal investigator.
- In-office email or fax.
- Willingness to follow the study protocol and to co-operate with the study monitors.

This clinical study is designed to be in conformance with the ethical principles in the Declaration of Helsinki, with the ICH guidelines for Good Clinical Practice (GCP) and all the applicable local guidelines.

## 6 Ethics Review / Statement of Compliance

#### 6.1 Relevant Standards / Guidelines

This implementation document has been developed in accordance with the following:

- ISO 14155. Clinical Investigation of Medical Devices
- ICH Harmonized Tripartite Guideline for Good Clinical Practice
- Declaration of Helsinki

#### 6.2 Institutional Review Board

This study was conducted in accordance with Institutional Review Board regulations (U.S. 21CFR Part 56.103) or applicable IEC regulations. Copies of all IRB/IEC correspondence with the investigator/sponsor will be kept on file. The study will commence upon approval from the following Institutional Review Board: Hospital Clínico San Carlos Profesor Martín Lagos, s/n. - Puerta G - 4ª Norte Madrid 28040 Madrid España. Tel. 91 330 34 13. Email. ceic.hcsc@salud.madrid.org.

### 6.3 Clinical Trial Registration

This study will be registered with clinical trials.gov in accordance with section 801 of the Food and Drug Administration (FDA) Act which mandates the registration of certain clinical trials of drugs and medical devices.

#### 6.4 Informed Consent

Informed consent, (Appendix 1), shall be obtained in writing from the subject and the process shall be documented before any procedure specific to the clinical investigation is carried out.

## 7 Potential Risks and Benefits to Human Subjects

There may be direct benefits to the subjects in this study such as improved vision, comfort, convenience, and cosmetic advantage. Participation in a study may contribute to scientific research information that may be used in the development of new contact lens products. In addition, subjects will receive an examination of the front part of their eyes and may have the opportunity to try a different type of soft contact lenses and/or different lens care products at no cost to them. The contact lens materials used in this study are commercially available intended for daily wear (NOT extended wear) similar to the average wearing time of 10-16 hours for daily wear lenses.

This study is considered to be a non-significant risk study based on United State Food and Drug administration (FDA) and International Standards Organization (ISO) guidelines because the study devices used as intended in this study (daily wear) don't represent a potential for serious risk to the health, safety or welfare of the subject, and (2) it is not an implant, (3) it is not used to support or sustain human life, (4) it is not of substantial importance in diagnosing, curing, mitigating or treating disease or otherwise prevents impairment of human health, (5) does not present a potential for serious risk to the health, safety or welfare of the subject.

Complications that may occur during the wearing of contact lenses include discomfort, dryness, aching or itching eyes, excessive tearing, discharge, hyperemia and variable or blurred vision. More serious risks may include photophobia, iritis, corneal edema or eye infection. Although contact lens-related infections are very infrequent, the possibility does exist. The incidence of infection due to day-wear soft lenses is 0.035%. Almost always an infection will occur only in one eye. This risk is assumed by 35-million Americans who currently wear contact lenses. Routine clinical procedures including auto-refraction, auto-keratometry, visual acuity, anterior ocular health assessment, and contact lens fitting will be used. In addition, high magnification imaging of the lens fit may be made using 35 mm or digital cameras, in vivo confocal microscopy, and/or specular microscopy. Patients will be monitored in the clinic during the study to reduce if not eliminate the occurrence of adverse or potential adverse events. Patients will be given instructions from the study investigator regarding early symptoms and signs of adverse events and their contact information.

## 8.1 Participants

Habitual soft toric contact lens wearers that provide written informed consent and meet the protocol entrance criteria. Subjects will be recruited from the investigator's private practice, Consultorio Optométrico, databases who agree to voluntarily participate in the study (Appendix 2, timeline). All subjects will be screened to determine study eligibility. Each subject will be given a unique ID number. Additionally, all subjects must meet the study inclusion and exclusion criteria listed below.

#### Inclusion criteria

A person is eligible for inclusion in the study if he/she:

- A person is eligible for inclusion in the study if he/she:
- Is between 18 and 40 years of age (inclusive)
- Has had a self-reported visual exam in the last two years
- Is an adapted soft contact lens wearer
- Is not a habitual wearer of either study lens
- Has a contact lens spherical prescription between plano to 10.00 (inclusive) best corrected visual acuity of 20/30 or better in either eye
- Have contact lens prescription of no less than -0.75D of astigmatism and no more than -1.75
   D in both eyes.
- Can achieve best corrected spectacle distance visual acuity of 20/25 (0.10 logMAR) or better in each eye.
- Can achieve a distance visual acuity of 20/30 (0.18 logMAR) or better in each eye with the study contact lenses.
- Has clear corneas and no active ocular disease
- Has read, understood and signed the information consent letter.
- Patient contact lens refraction should fit within the available parameters of the study lenses.
- Is willing to comply with the wear schedule (at least 5 days per week, > 8 hours/day assuming there are no contraindications for doing so).
- Is willing to comply with the visit schedule

#### **Exclusion Criteria**

A person will be excluded from the study if he/she:

- A person was excluded from the study if he/she:
- Has a CL prescription outside the range of the available parameters of the study lenses.
- Has a spectacle cylinder less than -0.75D or more than -1.75 D of cylinder in either eye.

- Has a history of not achieving comfortable CL wear (5 days per week; > 8 hours/day)
- Has contact lens best corrected distance vision worse than 20/25 (0.10 logMAR) in either eye.
- Presence of clinically significant (grade 2-4) anterior segment abnormalities
- Presence of ocular or systemic disease or need of medications which might interfere with contact lens wear.
- Slit lamp findings that would contraindicate contact lens wear such as:
  - Pathological dry eye or associated findings
  - o Pterygium, pinguecula, or corneal scars within the visual axis
  - Neovascularization > 0.75 mm in from of the limbus
  - o Giant papillary conjunctivitis (GCP) worse than grade 1
  - Anterior uveitis or iritis (past or present)
  - Seborrheic eczema, Seborrheic conjunctivitis
  - History of corneal ulcers or fungal infections
  - Poor personal hygiene
  - Has a known history of corneal hypoesthesia (reduced corneal sensitivity)
  - Has aphakia, keratoconus or a highly irregular cornea.
  - Has Presbyopia or has dependence on spectacles for near work over the contact lenses.
  - o Has undergone corneal refractive surgery.
  - Is participating in any other type of eye related clinical or research study.

## 8.2 Study Materials

#### 8.2.1 Contact lens

CooperVision will provide the site with an inventory of both study lenses (**LENS A**) and (**LENS B**) to allow participants to be fit with the lens powers available for this study.

All subjects will be trial fitted and, if suitable, dispensed the first pair of the assigned lens brand assigned per a determined table (Appendix 3). The lenses used in this study are all FDA approved and marketed products. Details of the study contact lenses are shown in Table 1.

Table1: Study lens parameters

| Brand | Biomedics 1 Day Toric<br>(LENS A) | MyDay Toric<br>(LENS B) |
|---|---|---|
| Manufacturer | CooperVision | CooperVision |
| Material | Ocufilcon D | stenfilcon A |
| FDA Class | Group 2 | Group 5 |
| WC % | 55% | 54% |
| Base Curve (mm) | 8.7 | 8.6 |
| Lens Diameter (mm) | 14.5 | 14.5 |
| Sphere Power (D) | Plano to -6.00D (0.25D steps)<br>-6.50D, -7.00D,<br>-7.50D to -10.00D | +8.00D to -10.00D (0.50D steps after +/- 6.00D) |
| Cyl Power (D) | -0.75, -1.25, -1.75 | -0.75, -1.25, -1.75 |
| Axis (degrees) | 180, 160, 90, 20 | Full circle in 10° steps |
| Wearing schedule | Daily disposable wear | Daily disposable wear |

#### 8.2.2 Contact Lens care

As this is a daily disposable study, no lens care will be required.

#### 8.2.3 Storage of Study Medications/Treatments

There are no unapproved investigational products used in this study requiring special storage accommodations.

#### 8.2.4 Clinical Supply Inventory

There are no unapproved investigational products used in this study requiring special inventory requirements.

#### 8.2.5 Disposal of Consumables

This study dispenses consumables (lenses) to participants for use during the study. Study lenses worn by participants will be discarded by the principal investigator at the end of the study.

#### 8.2.6 Masking and Control of Study Materials

The contact lenses, (**LENS A**, and **LENS B**), will be masked to the subject only. The lenses will be removed from their blister pack by an assistant and transferred to an unmarked lens case to maintain the participants masked of the study lenses. Participants will then be instructed to remove the lenses from the lens case and insert them onto their eyes. It is not possible for the study investigators to be

masked because of the need to follow the specific lens fitting guide during the lens prescription optimization visit.

### 8.2.7 Ordering and Accountability of Study Materials

The study sponsor will supply the investigators with the study lenses to use during the study.

#### 8.3 Visit Schedule and Procedures

This will be an interventional, subject masked, bilateral, non-dispensing fitting study. Participants will be examined at two different points over the course of one day, lens dispensing, and 15 minutes post lens settling. Participants will wear two different pairs of lenses with **LENS A** fitted first to all participants, followed by **LENS B**. Anterior ocular health examination will be performed at baseline without the use of fluorescein\*.

The following outline identifies the four study visits and the general procedures, (Appendix 5), to be conducted at each visit for each day of the study and recorded in the case report forms (Appendix 6):

#### 8.3.1 Visit 1: Baseline / Trial Fit / Lens order

- Subjects should attend this visit wearing their **spectacle** lenses
- Explanation of the study.
- Sign informed consent form.
- Collect habitual toric lens brand information
  - Brand
  - Power(s)
  - Replacement schedule (daily, 2-week, monthly)
- Anterior ocular health examination (Slit lamp without fluorescein).
- Insert trial toric LENS A, evaluate the fit and optimize the prescription if needed based on over-refraction.



Order final LENS B.

<sup>\*</sup> Fluorescein will not be used before lens dispensing to prevent potential eye discomfort that could influence subjective comfort ratings after lens fitting and settling. However, fluorescein will be instilled at the last visit upon lens removal.

## 8.3.2 Visit 2: Lens dispensing (Fit LENS A / Evaluate)

• Subjective assessments ➤ Handling on insertion (0 -100 scale). 8.3.3 Visit 3: 15 minutes (Evaluate LENS A) 8.3.4 Visit 3: Lens dispensing (Fit LENS B / Evaluate)

Subjective assessments

- ➤ Handling on insertion (0 -100 scale).
- > Comfort on insertion (0 -100 scale)



## 8.3.5 Visit 4: 15 minutes (Evaluate LENS B / Study Exit)



> Complete the study exit

## 9 Adverse Event Reporting

## 9.1 Adverse Response Definitions

**Adverse Event (AE)**: An AE refers to any untoward medical occurrence (sign, symptom or disease) in a trial subject that does not necessarily have a causal relationship with the study device. AEs may be classified as 'unanticipated adverse device effects,' 'serious AEs,' 'significant AEs,' or 'non-significant AEs,' as defined below.

| Classification | Definition |
|---|---|
| Serious<br>Adverse Event | Those events that are life-threatening, or result in permanent impairment of a body function, or permanent damage to a body structure or necessitate medical (therapeutic) or surgical intervention to preclude permanent impairment of a body function or permanent damage to a body structure. |
| Unanticipated Adverse Device Effect | Adverse events in a clinical trial that were not previously identified in the protocol in terms of nature, severity, or degree of incidence. An Unanticipated Serious Adverse Device Effect is an unanticipated adverse event that is serious in nature and caused by or associated with the device and is considered reportable. |
| Significant Adverse Event | Those non-serious adverse events that occur with contact lens usage that are not sight-threatening but are usually symptomatic and may warrant therapeutic management and /or temporary or permanent discontinuation of contact lens wear. |
| Non-Significant<br>Adverse<br>Events | Those less severe non-serious adverse events that occur with contact lens usage that are not sight-threatening, may or may not be symptomatic and may warrant palliative management, such as ocular lubricants or temporary interruption of contact lens wear. |

AE classification, coding (for reporting to the sponsor) and examples are provided in the following table of Contact LENS Adverse Event Classification and Reporting:

| Code | Condition | Potential AE<br>Classification | Reporting |
|---|---|---|---|
| 01 | Presumed infectious corneal ulcer | SERIOUS | |
| 02 | Permanent loss of ≥2 lines of best spectacle corrected visual acuity (BSCVA) | SERIOUS | |
| 03 | Corneal injury that results in permanent opacification within central cornea (6mm) | SERIOUS | Notify sponsor as |
| 04 | Neovascularization within the central 6mm of cornea | SERIOUS | soon as possible,<br>within 24 hrs; IRB |
| 05 | Uveitis or Iritis | SERIOUS | reporting as per |
| 06 | Endophthalmitis | SERIOUS | requirements |
| 07 | Hyphema | SERIOUS | |
| 08 | Hypopyon | SERIOUS | |
| 09 | Persistent epithelial defect | SERIOUS | |
| 00 | Other serious event | SERIOUS | |

| 11 | Peripheral non-infectious ulcer (outside central 6mm) | SIGNIFICANT | |
|---|---|---|---|
| 12 | Symptomatic corneal infiltrative events | SIGNIFICANT | |
| 13 | Superior epithelial arcuate lesions (SEALs) involving epithelial split | SIGNIFICANT | |
| 14 | Any temporary loss of ≥2 lines BSCVA for ≥2wks | SIGNIFICANT | |
| 15 | Corneal staining ≥ dense coalescent staining up to 2mm in diameter (i.e. moderate staining) | SIGNIFICANT | |
| 16 | Corneal neovascularization ≥ 1.0mm to 1.5mm vessel penetration (if 2 Grade change from baseline) | SIGNIFICANT | Notify sponsor as |
| 17 | Any sign and/or symptom for which subject is administered therapeutic treatment or which necessitates discontinuation of lens wear for ≥ 2 weeks | SIGNIFICANT | soon as possible,<br>within 5 working<br>days; IRB reporting<br>as per |
| 10 | Other significant event | SIGNIFICANT | requirements |
| 21 | Conjunctivitis: bacterial, viral, allergic | NON-SIGNIFICANT | |
| 22 | Papillary conjunctivitis if ≥ mild scattered papillae/follicles approximately 1mm in diameter (if 2 Grade change from baseline) | NON-SIGNIFICANT | |
| 25 | Asymptomatic corneal infiltrative events | NON-SIGNIFICANT | |
| 26 | Localized allergic reaction | NON-SIGNIFICANT | |
| 27 | Contact dermatitis | NON-SIGNIFICANT | |
| 28 | Any sign and/or symptom for which temporary lens discontinuation for > 1 day is recommended | NON-SIGNIFICANT | |
| 20 | Other non-significant sign and/or symptom | NON-SIGNIFICANT | |

#### Normal or adaptive symptoms

Transient symptoms such as end-of-day dryness, LENS Awareness, itching or burning or other discomfort may occur with contact lens wear and may occasionally reduce wearing time. These are not reported as adverse events unless they are unexpected in nature, severity or rate of occurrence.

#### 9.2 Procedures for Adverse Events

Treatment of an adverse event will depend on its nature and severity. Based on the clinical judgment of the investigator the subject may be referred to an ophthalmologist for treatment. The investigator will attempt to determine whether the reaction is related to the test device or a result of other factors. An Adverse Event Form will be completed for each adverse event. If both eyes are involved, a separate

Adverse Event Form will be completed for each eye. Whenever possible, the adverse event will be photo-documented.

Expenses incurred for medical treatment as part of study participation will be paid by the sponsor (bills and prescription receipts kept). The subject must be followed until resolution and a written report completed indicating the subsequent treatment and resolution of the condition.

## 9.3 Reporting Adverse Events

All potential **Serious and Unanticipated Adverse Device Effects** that are related or possibly related to subject participation in the investigation will be reported to the Principal Investigator and the sponsor within 24 hours of the investigator becoming aware of the event. The Principal Investigator will report the event to the EC/IRB as soon as possible (by fax, mail/delivery, phone, or email), but within 10 business days of becoming aware of the problem. *All fatal or life threatening events will be reported immediately to the IRB*.

**Significant and Non-Significant Adverse Events** will be reported to the sponsor as soon as possible, but no later than 5 working days after the occurrence.



## 9.4 Discontinuation from the Study

All discontinuations will be fully documented on the appropriate CRF Exit and Adverse Event forms as needed. Participants will be followed until resolution (in most instances) and are free of the ophthalmic insert related complications or other ocular pathology. When possible study lenses involved in an Adverse Event will be returned to the sponsor in a new tightly sealed contact lens case, and labeled with the subject identification and stored in Unisol non-preserved saline.

## 10 Statistical Analysis

## 10.1 Statistical analysis

Summary statistics will be produced, (e.g., mean, standard deviation), by the principal investigator. Differences between lenses will be compared using Paired t-tests. Paired t-tests /analysis of variance for normal (interval/continuous) data, Wilcoxon's signed ranks test for non-normal (ordinal) data, chi-squares test for nominal data. A Binomial test will be used to evaluate lens preference questions. All participants who are evaluated in the study will be used in the analysis. In the event of missing data individual number of points will be excluded in the analysis and not extrapolated from the collected Confidential

data. The critical alpha level for statistical significance will be set at  $p \le 0.05$ , with adjustment for multiple comparisons.

### 10.2 Sample size

Figure 1 shows the sample size calculation for a paired t-test, (alpha=0.05), in order to detect a difference in mean subjective handling scores between lenses. Assuming a standard deviation of 1.2, a sample size of about 37 completed subjects provides 84% power to detect a difference in subjective handling ratings of 0.6 points on a 0-10 scale. However, in this study a scale of 0-100 will be used. In order to account for potential subject dropouts or AEs, around 45 subjects will be enrolled with the aim to complete 37.

Figure 1. Sample size calculation (Minitab 20.2. Statistics software)





## 11.1 Study monitoring

A site visit or discussion may be conducted during the course of the study as appropriate. Prior to final data freeze, a close-out visit/discussion may be warranted to check for accuracy and completeness of records. The sponsor or sponsor's representatives will be authorized to gain access to the source documentation for the purposes of monitoring and auditing the study.

### 11.2 Record keeping

Detailed records of all study visits will be made using the Case Report Forms (CRFs).

#### 11.3 Record retention

Following study completion, data will be available in electronic and/or paper format for audit, sponsor use, or subsequent analysis. The original clinical raw data (including completed CRFs and Informed Consent forms) will be retained according to guidelines set forth in the general work agreement with the site. The Sponsor will be notified and consulted if ever the files are to be destroyed. In the event that this implementation document is indicated for design verification and validation purposes, as indicated on the title page, all original raw data forms and completed CRF's will be forwarded to the sponsor at completion of the final report.

## 11.4 Data Entry / Data Management

Data will be entered into an electronic spreadsheet. Study staff will only be able to modify the data file via password entry. The investigators will be responsible for the data integrity, and complete data entry for each visit as well as the take home questionnaires. The investigator will send the data collected to the study sponsor within 5 business days after the last subject completes the final visit. A full report will be provided by the investigator at the mutually agreed timeline after the study completion date.

## 11.5 Confidentiality

This study is confidential in nature. All information gathered during this study is proprietary and should be made available only to those directly involved in the study. Information and reports arising from this project are the property of the sponsor.

In accordance with the provisions of Regulation (EU) 2016/679 of the European Parliament and of the Council, of 27 April 2016 (General Data Protection Regulation) and Organic Law 3/2018, on Personal Data Protection and guarantee of digital rights, all data collected here will be incorporated into a file called "Datos Pacientes" (Patient Data), whose responsible is the principal investigator and protected under username and password. The paper file will be kept under lock and key in the Management Office of the University Optometry Clinic of the Faculty of Optics of the Complutense University of Madrid. The interested participant may exercise his/her rights of access, rectification, cancellation and opposition by writing to the principal investigator (Juan Gonzalo Carracedo Rodríguez, Facultad de Óptica y Optometría, C/ Arcos de Jalón 118, 28037 Madrid).

#### 11.6 Publication

The investigators will not be permitted to publish or present at scientific meetings results obtained from the clinical study without prior written consent from the sponsor.

## 12 Study Costs and Subject Compensation

CVI will compensate the Investigator, (principal investigator), and the Subjects, (each a "Subject" and together the "Subjects"), for their time and participation in this voluntary study. Payments to the Clinical Investigator are per subject visit with a total of 4 visits for 37- 45 subjects. The study lenses will be provided by the sponsor to the Clinic Site. Clinical Site will receive the payment for the Subjects and are responsible in distributing the subject's compensation.

Complete outline/details of the payment compensation are detailed in the Clinical Study Agreement. The statistical analysis, and study final report are "one-time costs" There will be no payments to the Clinical Site for interim visits, unless Subjects are visiting regarding an adverse event. Data from interim office visits, if mandated by your clinic, can be collected and entered using the unscheduled visit form.

Expenses incurred for medical treatment as part of Study participation will be paid by CVI (bills and prescription receipts kept). The Subject must be followed until resolution and a written report is completed indicating the subsequent treatment and resolution of the condition.